CLINICAL TRIAL: NCT02834494
Title: 3D Elastography (Shear Wave) : Assessment of Response to Neo-adjuvant Chemotherapy (NACT) : in Vivo Quantification, for Patients With a Locally Advanced Breast Cancer.
Brief Title: Assessment of Response to Neo-adjuvant Chemotherapy for Patients With a Locally Advanced Breast Cancer With 3D Elastography (Shear Wave), NEOELASTO
Acronym: NEO-ELASTO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IC 2015-07
Record Dates: First submitted 2016-07-08; First posted 2016-07-15 (Estimated); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Breast Neoplasms
Keywords: locally advanced breast cancer; neoadjuvant chemotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 3D Shear Wave Elastography (SWE) (Other)
  Interventions: Procedure: 3D Shear Wave Elastography (SWE); Biological: Biopsy

INTERVENTIONS:
Procedure: 3D Shear Wave Elastography (SWE) — Ultrasound imaging with Elastography will be performed at the inclusion (T0), after course 1 and course 2 respectively with anthracyclines, at the end of anthracycline treatment and at the end of taxane treatment.
Biological: Biopsy — Optional biopsy of breast tumor under neoadjuvant chemotherapy after the course 2 of anthracycline.

SUMMARY:
Assess the accuracy of the sequential measurements by 3D Shear Wave Elastography (SWE) for predicting histological response to neoadjuvant chemotherapy in patients with locally advanced breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Infiltrating Breast Cancer untreated and/or locally advanced (stages I (T1c), IIa IIb, IIIa, IIIb, IIIc of UICC classification), whatever histological type.
* Neo-adjuvant chemotherapy decided.(Anthracyclines, taxanes and, for tumors overexpressing human epidermal growth factor receptor 2 (HER2) protein, targeted recombinant humanized monoclonal antibodies)
* Index tumor whose dimensions are between 10 to 50 mm. Multifocality, and/or multicentricity and/or bilaterality accepted (maximum 2 tumors by breast et tumors well differentiated from each other).
* Patients aged at least 18 years old at diagnosis
* Full results conventional breast exams available and no reason to achieve MRI breast exam
* Patient explanation given and consent information signed

Exclusion Criteria:

* Pregnant or during lactation
* Personal history of ipsilateral breast cancer (ipsilateral recurrence or second cancer in the same breast).
* Patient carrier of cosmetic breast implants
* Person deprived of liberty or under guardianship
* Contraindication for receiving neo-adjuvant chemotherapy for any medical reason
* Inability to submit to medical monitoring of the trial for reasons of geography, social or psychological.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2016-02-22 (Actual); Primary Completion 2020-09-09 (Actual); Study Completion 2020-09-09 (Actual)

PRIMARY OUTCOMES:
Assess the accuracy of the sequential measurements by 3D Shear Wave Elastography (SWE) for predicting histological response to neoadjuvant chemotherapy | up to 32 months
  Measure of the tumor prior to neoadjuvant chemotherapy (T0), at T1 and T2(1stand 2nd courses of anthracycline), at mid-treatment between anthracycline and taxane chemotherapy (Tmi), at the end of chemotherapy before surgery (Tfin).

SECONDARY OUTCOMES:
Elastic properties before treatment (especially ratio between tumor and glandular breast or fat tissues close to the tumors) | up to 32 months
  Use technic Supersonic Shear Imaging.
peritumoral environmental elasticity properties | up to 32 months
  Use technic Supersonic Shear Imaging (Explorer, Supersonic Imagine).
Reliable early biomarker of histological response. | up to 32 months
  Estimate under chemotherapy if early changes in tumor's elasticity can provide a reliable early biomarker of histological response.
tumor volume changes under treatment by 3D ultrasound | up to 32 months
  Estimate tumor volume changes under treatment by 3D ultrasound and Compare with measurements obtained by other conventional imaging methods currently used for monitoring patients under neoadjuvant chemotherapy
Compare changes in tumor elasticity under chemotherapy to variables obtained by other imaging modalities (Breast MRI) performed in clinical routine | up to 32 months
Compare changes in tumor elasticity under neoadjuvant chemotherapy to changes in diffusion apparent coefficient by using technic Supersonic Shear Imaging (Explorer, Supersonic Imagine). | up to 32 months
Compare changes in tumor volume to histological response (Gold Standard : surgery after neoadjuvant chemotherapy according to " Residual Cancer Burden " score | up to 32 months
Compare predictive value (semi-quantitative et quantitative measurements) of tumor elasticity | up to 32 months
Assess vascular shape and its evolution under treatment by Ultrasensitive Doppler technic "Ultra-Fast Doppler" | up to 32 months
Compare tumor elasticity to conventional histological parameters | 6 weeks
  For the additional biopsy (optional) under neoadjuvant chemotherapy at T2, correlation elastography to pathological parameters of peritumoral environment by analyzing conventional histological parameters.

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Curie Paris, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Sponsor will share de-identified data sets. Documents generated under the project will be disseminated in accordance with Institut Curie policies.
Supporting Information: SAP
Time Frame: Data requests can be submitted starting 9 months after last article publication and will be made accessible for up to 12 months.
Access Criteria: Access to trial individual participant data can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a data sharing agreement (DSA).